CLINICAL TRIAL: NCT05127902
Title: Association Between Postural Balance and Muscle Activity of the Lumbar and Lower Limb Muscles in Female With or Without Adolescent Idiopathic Scoliosis (AIS) During Standing Balance Tasks With Upper Limb Movement
Status: Completed | Type: Observational
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Chak Long Hay Forest, Principal Investigator, Tung Wah College
Other Study IDs: MHS_SRC_2021_010
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adolescent idiopathic scoliosis group: Female subjects aged 10 to 16 will be recruited if they are diagnosed with AIS by standard standing long X-ray examinations, with Cobb angle larger or equal to 15°, without prior treatment for their AIS and been cleared for physical activity by their doctors. Subjects were excluded if they had (i) Cobb angle larger or equal to 40°, (ii) scoliosis with any known aetiologies such as congenital, neuromuscular, metabolic, and skeletal dysplasia, (iii) known endocrine and connective tissue abnormalities, (iv) known heart condition or other diseases that could affect the safety of exercise, (v) eating disorders or gastrointestinal malabsorption disorders, and (vi) currently taking medications that affecting their bone or muscle metabolism. All subjects will be recruited in the community.
  Interventions: Diagnostic Test: Proprioceptive-stabilometric assessment machine (ProKin 252, TecnoBody®, Italy)
- Control group: Ten healthy female subjects with matched for age, height and weight will be recruited as control.
  Interventions: Diagnostic Test: Proprioceptive-stabilometric assessment machine (ProKin 252, TecnoBody®, Italy)

INTERVENTIONS:
Diagnostic Test: Proprioceptive-stabilometric assessment machine (ProKin 252, TecnoBody®, Italy) — Proprioceptive-stabilometric assessment machine (ProKin 252, TecnoBody®, Italy) Balance performance of subjects will be tested on the proprioceptive-stabilometric assessment machine.
  Noraxon wireless TELEmyo Direct Transmission System (TELEmyo DTS) with product code of 580 (Noraxon, USA Inc., USA)
  The sampling frequency will be of 1000Hz and bandwidth of 10-500Hz. Bipolar silver chloride electrodes of 15mm diameter will be used for EMG signals collection, the interelectrode distance will be fixed at 20mm. Normalization procedure will be done by asking subjects to perform isometric maximum voluntary contractions (MVC). The MVC will be measured by Lafayette hand-held dynamometer connected to flat stirrup. MVC will be tested as listed below.
  The sEMG signals during each experiment will be normalized to the sEMG at isometric MVC and expressed as percentages of the maximum sEMG activity (%EMG_max) for comparison with normalization signal processing program in Noraxon System.
  Other Names: Noraxon wireless TELEmyo Direct Transmission System (TELEmyo DTS) with product code of 580 (Noraxon, USA Inc., USA)

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is the most common type of three-dimensional deformity of the spine in adolescence with a clear female predominance at a prevalence rate of 3.5% in Hong Kong. AIS increases the risk of spinal degeneration, back pain, and cardiorespiratory dysfunction. These impairments caused by AIS can be related to the abnormal lateral deviation, axial rotation, and reduction of sagittal curves of the spine. AIS has been associated with asymmetrical muscle activity and impaired postural balance performance. AIS who had convex side of the major curves to the right demonstrated an increase in right side thoracic and lumbar erector spinae muscle activity during pelvic anterior, posterior, and left tilting on an unstable sitting board as measured by electromyography (EMG).

Postural balance is defined as the act of maintaining, achieving and restoring a state of balance during any posture or activity. The ability of maintaining postural balance in AIS is influenced by multiple factors including spinal deformities, asymmetrical muscle activities, alteration in sensory input, central integration or motor response. Previous studies have investigated the motor response in young adults. They were found to depend more on ankle strategy than hip strategy during a balance perturbation on a movable platform. Increased lateral gastrocnemius muscle activity was also observed when centre of gravity falls forward during an EMG measurement in quiet stance. In a study of low back pain patients, training regime involving single rapid arm movement in flexion and extension was found to promote the activation of the transversus abdominis muscle and improved the feedforward postural adjustment. There are limited studies to investigate the association between somatosensory input and motor response particularly lower limb muscle activity and upper limb movement on balance control in AIS. Recent evidence also suggested that AIS tend to overestimate the severity of their spinal deformity but their perception of their body schema and spinal curvature can be improved by enhancing motor skills. Therefore, training of postural balance that involved enhancing motor skills and stimulating somatosensory system will have the potential to improve motor response as well as improve self-perceived body schema in AIS.

DETAILED DESCRIPTION:
Ten female subjects aged 10 to 16 will be recruited if they are diagnosed with AIS by standard standing long X-ray examinations, with Cobb angle larger or equal to 15°, without prior treatment for their AIS and been cleared for physical activity by their doctors. Subjects were excluded if they had (i) Cobb angle larger or equal to 40°, (ii) scoliosis with any known aetiologies such as congenital, neuromuscular, metabolic, and skeletal dysplasia, (iii) known endocrine and connective tissue abnormalities, (iv) known heart condition or other diseases that could affect the safety of exercise, (v) eating disorders or gastrointestinal malabsorption disorders, and (vi) currently taking medications that affecting their bone or muscle metabolism. Ten healthy female subjects with matched for age, height and weight will be recruited as control. All subjects will be recruited in the community.

All subjects will participate voluntarily in this study. Informed consent will be signed by subject in the presence of their parents after thorough explanation by research personnel before data collection. This study will be carried out with Low/Negligible Risk Human Research Ethics Approval issued by TWC Research Ethics Committee (REC).

Study Procedures This cross-sectional study will be carried out at Physiotherapy laboratory, School of Medical and Health Sciences, Tung Wah College between October 2021 and May 2022.

The experiment environment will be maintained at 25 degrees Celsius. Subjects should not perform any vigorous exercise before testing time.

Subjects will be asked to complete 3 questionnaires: The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY), Tanner Scale and Trunk Appearance Perception Scale (TAPS) prior to the experiment for determining their physical activity level, sexual maturity and self-perception of spinal deformity respectively. Bioelectric Impedance Analysis (BIA) will be done to collect body composition data. Anthropometric parameters and spinal deformity data will be collected by female student investigators.

Surface EMG (sEMG) electrodes will be used for detection of muscle activity during balance tasks. According to the Surface EMG for Non-Invasive Assessment of Muscles (SENIAM) guidelines, skin preparation with hair removal by single-use razor and alcohol swab will be done before applying electrodes to reduce the skin impedance below 5k Ohm. sEMG electrodes will be positioned on muscle bellies of erector spinae (ES) at lumbar level (largest muscle mass lateral to L3 spinous process). For gluteus medius (GM), electrodes will be placed at proximal 1/3 of the distance between iliac crest and the greater trochanter. For lateral gastrocnemius (LG), electrodes will be placed at most prominent part of muscle belly during resisted plantar flexion.

After placing the sEMG for muscle activity measurement, balance performance of subjects will be tested on a proprioceptive-stabilometric assessment machine. Four tasks will be carried out, including: 1) open eyes fixing at a set point (170 cm height and 200 cm away) on a wall with relaxed arm aside; 2) eyes closed with relaxed arm aside; 3) eyes open with arm movements and 4) eye closed with arm movements. The arm movements are unilateral shoulder flexion and and extension of both arms with two frequencies (40 bpm and 120 bpm). The tempo will be given using a metronome. Each task will be tested twice with at least fifteen seconds rest between trials.

Balance Functions Performance for each balance test will be recorded by proprioceptive-stabilometric assessment machine (ProKin 252, TecnoBody®, Italy). The outcome will be analysed in terms of Ellipse area (mm2), Perimeter (mm), Forward-backward standard deviation (mm), Medial-lateral standard deviation, Average center of pressure in the medial-lateral direction on X-axis projection (mm), Average center of pressure in the anterior-posterior direction on Y-axis projection (mm), Standard deviation of forward-backward displacement (mm), Standard deviation of medial-lateral displacement (mm), Average velocity for forward-backward displacement (mm/s), Average velocity for medial-lateral displacement (mm/s) and Standard deviation of Trunk sway (o).

sEMG Muscle Activity The muscle activity will be measured by surface electromyography and recorded by the Noraxon wireless TELEmyo Direct Transmission System (TELEmyo DTS) with product code of 580 (Noraxon, USA Inc., USA). The sampling frequency will be of 1000Hz and bandwidth of 10-500Hz. Bipolar silver chloride electrodes of 15mm diameter will be used for EMG signals collection, the interelectrode distance will be fixed at 20mm. Electrodes will be attached to surface of 3 groups of muscles bilaterally, namely the lumbar erector spinae (LES), gluteus medius (GM) and lateral gastrocnemius (LG). Placement of electrodes will be based on previous studies to reduce inconsistency and inter-subject variability in normalizing the sEMG signal [21]. Normalization procedure will be done by asking subjects to perform isometric maximum voluntary contractions (MVC). The MVC will be measured by Lafayette hand-held dynamometer connected to flat stirrup. MVC will be tested as listed below. For LES, resisted lumbar extension against belt on lower thoracic area (T12) in prone lying. For GM, resisted hip abduction against belt in side-lying. For LG, resisted ankle plantarflexion in sitting position against belt in 90º dorsiflexion.

The sEMG signals during each experiment will be normalized to the sEMG at isometric MVC and expressed as percentages of the maximum sEMG activity (%EMG_max) for comparison with normalization signal processing program in Noraxon System.

ELIGIBILITY:
Inclusion Criteria:

(i) Cobb angle larger or equal to 40° (ii) scoliosis with any known aetiologies such as congenital, neuromuscular, metabolic, and skeletal dysplasia (iii) known endocrine and connective tissue abnormalities (iv) known heart condition or other diseases that could affect the safety of exercise (v) eating disorders or gastrointestinal malabsorption disorders (vi) currently taking medications that affecting their bone or muscle metabolism

Exclusion Criteria:

-

Ages: 10 Years to 16 Years | Sex: Female
Age Groups: Child
Study Population: Recruited from community
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Balance function | 1 hour
  Ellipse area (mm2), Perimeter (mm), Forward-backward standard deviation (mm), Medial-lateral standard deviation, Average center of pressure in the medial-lateral direction on X-axis projection (mm), Average center of pressure in the anterior-posterior direction on Y-axis projection (mm), Standard deviation of forward-backward displacement (mm), Standard deviation of medial-lateral displacement (mm), Average velocity for forward-backward displacement (mm/s), Average velocity for medial-lateral displacement (mm/s) and Standard deviation of Trunk sway (o).
sEMG Muscle Activity | 1 hour

SECONDARY OUTCOMES:
Angle of trunk rotation (ATR) | 10 minutes
Anthropometric Measurements | 5 minutes
  Standing height, Sitting height and Arm span
Body composition | 5 minutes
  body fat mass (BFM), fat-free mass (FFM), body fat percentage (%BFM) and visceral adipose tissue (VAT), BMI
Sexual Maturity | 5 minutes
  Puberty maturity level including age of menarche correct to nearest month, breast development and pubic hair distribution will be self-assessed by subjects using Tanner Scale
Physical Activity Level | 5 minutes
  self-administered, 1-item questionnaire that measures the physical activity level with the consideration of frequency, duration, and intensity of the physical activity. CUHK-PARCY results in a score that stratifies subjects as low, moderate, and high in physical activity.
Self-perceived Spinal Appearance | 5 minutes
  the Trunk Appearance Perception Scale (TAPS) includes 3 sets of figures from 3 viewpoints: looking toward the back, looking toward the head with the patient bending over (Adam's test), and looking toward the front. Each drawing is scored from 1 (greatest deformity) to 5 (smallest deformity) and a mean score is obtained by adding the scores for the 3 drawings and dividing by 3

CONTACTS AND LOCATIONS:
Locations (1):
- Tung Wah College, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The possible IPD to be shared include the primary outcome measure and secondary outcome measure.

REFERENCES:
- [Background] Fong DY, Cheung KM, Wong YW, Wan YY, Lee CF, Lam TP, Cheng JC, Ng BK, Luk KD. A population-based cohort study of 394,401 children followed for 10 years exhibits sustained effectiveness of scoliosis screening. Spine J. 2015 May 1;15(5):825-33. doi: 10.1016/j.spinee.2015.01.019. Epub 2015 Jan 20. PMID 25615844
- [Background] Nishida M, Nagura T, Fujita N, Hosogane N, Tsuji T, Nakamura M, Matsumoto M, Watanabe K. Position of the major curve influences asymmetrical trunk kinematics during gait in adolescent idiopathic scoliosis. Gait Posture. 2017 Jan;51:142-148. doi: 10.1016/j.gaitpost.2016.10.004. Epub 2016 Oct 11. PMID 27764749
- [Background] Smania N, Picelli A, Romano M, Negrini S. Neurophysiological basis of rehabilitation of adolescent idiopathic scoliosis. Disabil Rehabil. 2008;30(10):763-71. doi: 10.1080/17483100801921311. PMID 18432434
- [Background] Cheung J, Veldhuizen AG, Halberts JP, Sluiter WJ, Van Horn JR. Geometric and electromyographic assessments in the evaluation of curve progression in idiopathic scoliosis. Spine (Phila Pa 1976). 2006 Feb 1;31(3):322-9. doi: 10.1097/01.brs.0000197155.68983.d8. PMID 16449906
- [Background] Jung JY, Cha EJ, Kim KA, Won Y, Bok SK, Kim BO, Kim JJ. Influence of pelvic asymmetry and idiopathic scoliosis in adolescents on postural balance during sitting. Biomed Mater Eng. 2015;26 Suppl 1:S601-10. doi: 10.3233/BME-151351. PMID 26406054
- [Background] Pasha S, Baldwin K. Are we simplifying balance evaluation in adolescent idiopathic scoliosis? Clin Biomech (Bristol). 2018 Jan;51:91-98. doi: 10.1016/j.clinbiomech.2017.11.011. Epub 2017 Nov 29. PMID 29277028
- [Background] Sahlstrand T, Ortengren R, Nachemson A. Postural equilibrium in adolescent idiopathic scoliosis. Acta Orthop Scand. 1978 Aug;49(4):354-65. doi: 10.3109/17453677809050088. PMID 696275
- [Background] Le Berre M, Guyot MA, Agnani O, Bourdeauducq I, Versyp MC, Donze C, Thevenon A, Catanzariti JF. Clinical balance tests, proprioceptive system and adolescent idiopathic scoliosis. Eur Spine J. 2017 Jun;26(6):1638-1644. doi: 10.1007/s00586-016-4802-z. Epub 2016 Nov 14. PMID 27844226
- [Background] Byl NN, Gray JM. Complex balance reactions in different sensory conditions: adolescents with and without idiopathic scoliosis. J Orthop Res. 1993 Mar;11(2):215-27. doi: 10.1002/jor.1100110209. PMID 8483034
- [Background] Pollock AS, Durward BR, Rowe PJ, Paul JP. What is balance? Clin Rehabil. 2000 Aug;14(4):402-6. doi: 10.1191/0269215500cr342oa. PMID 10945424
- [Background] Gatev P, Thomas S, Kepple T, Hallett M. Feedforward ankle strategy of balance during quiet stance in adults. J Physiol. 1999 Feb 1;514 ( Pt 3)(Pt 3):915-28. doi: 10.1111/j.1469-7793.1999.915ad.x. PMID 9882761
- [Background] Tsao H, Hodges PW. Persistence of improvements in postural strategies following motor control training in people with recurrent low back pain. J Electromyogr Kinesiol. 2008 Aug;18(4):559-67. doi: 10.1016/j.jelekin.2006.10.012. Epub 2007 Mar 2. PMID 17336546
- [Background] Notarnicola A, Farì G, Maccagnano G, Riondino A, Covelli I, Bianchi FP, et al. Teenagers' perceptions of their scoliotic curves. An observational study of comparison between sports people and non-sports people. Muscle Ligaments Tendons J 2019;09:225-35. https://doi.org/10.32098/mltj.02.2019.11
- [Background] Kong AP, Choi KC, Li AM, Hui SS, Chan MH, Wing YK, Ma RC, Lam CW, Lau JT, So WY, Ko GT, Chan JC. Association between physical activity and cardiovascular risk in Chinese youth independent of age and pubertal stage. BMC Public Health. 2010 Jun 3;10:303. doi: 10.1186/1471-2458-10-303. PMID 20525239
- [Background] Chan NP, Sung RY, Kong AP, Goggins WB, So HK, Nelson EA. Reliability of pubertal self-assessment in Hong Kong Chinese children. J Paediatr Child Health. 2008 Jun;44(6):353-8. doi: 10.1111/j.1440-1754.2008.01311.x. PMID 18476928
- [Background] Bago J, Sanchez-Raya J, Perez-Grueso FJ, Climent JM. The Trunk Appearance Perception Scale (TAPS): a new tool to evaluate subjective impression of trunk deformity in patients with idiopathic scoliosis. Scoliosis. 2010 Mar 25;5:6. doi: 10.1186/1748-7161-5-6. PMID 20338048
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Criswell E. Cram's Introduction to Surface Electromyography. 2nd ed. Sudbury: Jones and Bartlett Publishers; 2011.
- [Background] Cibulka M, Wenthe A, Boyle Z, Callier D, Schwerdt A, Jarman D, Strube MJ. VARIATION IN MEDIAL AND LATERAL GASTROCNEMIUS MUSCLE ACTIVITY WITH FOOT POSITION. Int J Sports Phys Ther. 2017 Apr;12(2):233-241. PMID 28515978
- [Background] Mochizuki G, Ivanova TD, Garland SJ. Postural muscle activity during bilateral and unilateral arm movements at different speeds. Exp Brain Res. 2004 Apr;155(3):352-61. doi: 10.1007/s00221-003-1732-x. Epub 2003 Dec 6. PMID 14661120
- [Background] Nairn BC, Drake JD. Impact of lumbar spine posture on thoracic spine motion and muscle activation patterns. Hum Mov Sci. 2014 Oct;37:1-11. doi: 10.1016/j.humov.2014.06.003. Epub 2014 Jul 12. PMID 25026559
- [Background] Sahli S, Rebai H, Ghroubi S, Yahia A, Guermazi M, Elleuch MH. The effects of backpack load and carrying method on the balance of adolescent idiopathic scoliosis subjects. Spine J. 2013 Dec;13(12):1835-42. doi: 10.1016/j.spinee.2013.06.023. Epub 2013 Oct 2. PMID 24095102
- [Background] Romano M, Minozzi S, Bettany-Saltikov J, Zaina F, Chockalingam N, Kotwicki T, Maier-Hennes A, Negrini S. Exercises for adolescent idiopathic scoliosis. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007837. doi: 10.1002/14651858.CD007837.pub2. PMID 22895967